CLINICAL TRIAL: NCT04371757
Title: Influence of the Autonomic Nervous System on Endothelial Function as an Acute Response to Exercise in Hypertensive Individuals: a Randomized Double-blind Protocol Study
Brief Title: Influence of the Autonomic Nervous System in Response to Exercise in Hypertensive Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Autonomic nervous system
Record Dates: First submitted 2020-04-16; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Autonomic Nervous System; Hypertension
Keywords: Endothelium; Physical Exercise
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Doxazosin; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomization for exercise interventions, as well as placebo or α1-adrenergic, will be performed using a computer program containing the coded distribution. The randomization of the subjects will be characterized as simple and divided into two parts; (A) directed to the three arms of exercise (aerobica exercise, resistido exercise and combinade exercise) and (B) the order in relation to the placebo or α1-adrenergic block.
Who Masked: Participant, Investigator
Masking Description: The allocation secrecy will be maintained until the time of the experiments, through a randomization list, in a remote place and without direct access by the researchers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercise session (Experimental): The aerobic exercise session will be performed on a horizontal cycle ergometer. A warm-up will be performed (5 minutes), followed by 40 minutes with moderate intensity (60% HRreserve) and controlled by a heart rate monitor, as well as the subjective effort scale (Borg 6 to 20 points). Blood pressure, heart rate and the Borg scale will be assessed at the beginning of aerobic exercise and every 5 minutes until the end.
  Interventions: Drug: α1-adrenergic block; Other: Placebo
- Resistance exercise session (Experimental): The resistance exercise session will be structured with knee extension, knee flexion, leg pressure and plantar flexion, in a station with guided weights, with 4x12 repetitions and 60% intensity of 1-RM; the cadence will be adjusted to 2:2 (concentric: eccentric) and controlled by a metronome. The rest between sets and exercises will be 90 seconds (total duration: 40 minutes). Blood pressure, heart rate and Borg scale will be recorded at the beginning and at the end of the 4th series of each exercise.
  Interventions: Drug: α1-adrenergic block; Other: Placebo
- Combined exercise session (Experimental): The combined exercise session will be structured with 20 minutes of resistance exercise + 20 minutes of aerobic exercise, as already described, except that the resistance exercises will have 2 sets of each exercise. As with other sessions, blood pressure, heart rate and the Borg scale will be assessed at the beginning and end of the second series of resistance exercise, as well as at the beginning and every 5 minutes of aerobic exercise up to 15 minutes after end of exercises.
  Interventions: Drug: α1-adrenergic block; Other: Placebo

INTERVENTIONS:
Drug: α1-adrenergic block — Ninety minutes before starting the experimental exercise protocol, participants will be offered a capsule containing an α-1 adrenoreceptor blocker (Drozazosin; 0.05 mg / kg-1 body weight) and will be instructed to lie down. All capsules will be handled by a specialized pharmacy.
  Other Names: Doxazosin
Other: Placebo — Ninety minutes before starting the experimental exercise protocol, participants will be offered a capsule containing an placebo (microcrystalline cellulose; 0.05 mg.kg-1 body weight) and will be instructed to lie down. All capsules will be handled by a specialized pharmacy.
  Other Names: Microcrystalline cellulose

SUMMARY:
Systemic arterial hypertension (SAH) has a direct association with endothelial dysfunction and major cardiovascular events. Evidence points to possible benefits of aerobic training in the endothelial function analyzed by the flow mediated dilation technique (flow mediated dilatation - FMD) in individuals with SAH. However, little is known about the influence of the autonomic nervous system (ANS) on the results of brachial artery FMD after different types of acute exercise in individuals with SAH. Thus, the objective of the research is to analyze the influence of the ANS on the FMD of the brachial artery of individuals with SAH after a session of aerobic (EA), resistance (ER) and combined (EC) exercise. For this, thirty-nine hypertensive individuals aged 35 to 55 years will be recruited and will be randomized to 2 sessions of AS, ER or EC. Also, within each modality, they will be randomized to α1-adrenergic block (Doxazosin 0.05 mg / kg-1) or placebo. The FMD will be performed by ultrasound 10 minutes before, as well as 10, 40 and 70 minutes after the exercise sessions and the autonomic control will be monitored (Finometer) for 10 minutes before each FMD. Arterial stiffness will also be analyzed, using the pulse wave velocity (PWV) by the Complior Analyzer. It is expected to demonstrate with this research the influence of the ANS on the FMD of the brachial artery in individuals with SAH in different physical exercises. This knowledge contributes to a better training prescription in this population.

DETAILED DESCRIPTION:
INTRODUCTION

Endothelial dysfunction precedes atherosclerosis. Endothelial cells play an important role in the modulation of vascular angiogenesis, inflammatory responses, homeostasis, as well as vascular tone and permeability. This vascular protection function is largely attributed to nitric oxide synthase endothelial, an enzyme responsible for the production of nitric oxide (NO).

The decrease in local NO bioavailability and/or insufficient vasomotor response characterizes endothelial dysfunction; a fact evidenced in situations such as SAH, diabetes mellitus, obesity, dyslipidemia, menopause and sedentary lifestyle. The evaluation of flow-mediated dilation (FMD) of the brachial artery, although it is an indirect method to assess endothelial function, is not invasive and a large part of its result depends on NO. The findings resulting from the acute stimulus of physical exercise can also predict long-term adaptations, therefore, it has been widely used.

Within this scenario, the change in lifestyle, including regular physical exercise, is part of the recommendations of antihypertensive therapy. The most cited factors, responsible for the potential antihypertensive effect and better endothelial response to long-term exercise include reduced sympathetic activity, balance between vasodilator and vasoconstrictor factors and reduced levels of vasoconstrictor endothelin-1.

Analyzes of a resistance exercise session in the FMD demonstrated that the knee extension exercise performed with moderate intensity, as well as, with light intensity can reduce the FMD 10-30-60 minutes after the session in individuals healthy. Interestingly, the same session, when performed at high intensity, was not able to provide changes in the FMD, leading to the idea of an inverse relationship between intensity of resistance exercise and FMD response. Recently, the investigators demonstrated that an aerobic exercise session, resisted and combined (resisted and aerobic) performed in moderate intensity for 40 minutes and exclusively with lower limbs, were not able to alter the FMD of the brachial artery of individuals with SAH when analyzed 10-40-70 minutes after the sessions. These results were accompanied by maintenance of endothelial microvesicle levels and factors involved with oxidative stress. Collectively, the investigators can raise the hypothesis that other factors, such as exacerbation of sympathetic activity in untrained members, may cause vasoconstriction and redirect blood flow to trained members, consequently, competing with endothelium-dependent vasodilating activity.

Researchers have shown that α1-adrenergic blockade with Phentolamine mitigated the reduction in blood flow in the forearm, demonstrated in a placebo condition, during a manual pressure exercise session in individuals with heart failure. Still, considering that the exacerbated activation of the sympathetic nervous system has been proposed as an important factor in the development and maintenance of SAH, the investigators can hypothesize that, after a session of acute physical exercise, there is a competition between the sympathetic activity (potentiating vasoconstriction) and endothelium-dependent vasodilation capacity, in individuals with SAH.

Whereas the acute effect of different modalities of physical exercise on FMD has conflicting results in healthy and hypertensive individuals, as well as a lack of information in the hypertensive population regarding the influence of SNA activity on vessel reactivity in response to physical exercise, the investigators developed a randomized clinical trial with the primary objective of analyzing the influence of autonomic nervous system activity on the FMD of the brachial artery of individuals with SAH after acute aerobic, resisted and combined (resisted and aerobic) exercise performed exclusively with lower limbs.

METHODS

Study setting.

The study will be carried out at the Institute of Cardiology of Rio Grande do Sul/Fundação Universitária de Cardiologia under the approval of the Ethics Committee of this Institution (UP 5678/19).

Eligibility criteria.

Men and woman with SAH, between 35-55 years old who attend the services of the Institute of Cardiology of Rio Grande do Sul and do not perform regular physical exercise (≥2 sessions per week) will be selected. The sample will exclude individuals with diabetes mellitus, chronic renal failure, body mass index (BMI) ≥35kg/m2, coronary artery disease, heart failure, not to be taking antihypertensive medication, making use of beta-blocker and/or alpha-blocker, present lesions in the lower limbs that prevent the protocol, smoking and menopause (woman).

Sample size.

Researchers have compared the FMD in healthy individuals after a session of aerobic exercise performed with the condition of placebo (SD 1.13%) and α1-adrenergic block (SD 1.91%) (difference of means: 3.1%). Thus, to find a similar difference in FMD between conditions (placebo and α1-adrenergic block) after our exercise session, the investigadors calculated a total sample of 15 individuals (α=0.05 and 80% power). For the comparison in FMD between the types of exercises, the pre-exercise (SD 1.18%) and post-exercise (SD 1.91%) of the α1-adrenergic block group. To find a difference in the FMD of 1.62% (α=0.05, power 80%), the calculated total sample was 30 individuals. Assuming a loss of 30% during the protocols, the total sample was 39 individuals.

Evaluation and interventions.

The volunteers will be selected from the information described in the medical records of the IC/FUC cardiology service. The first contact with the volunteer will be made via telephone in an attempt to check, a priori, the exclusion criteria.

Step 1. The individual's first visit to the IC/FUC will take place at the Clinical Research Laboratory (LIC) and all inclusion/exclusion criteria will be resumed. After the respective signature of the Informed Consent Form, the individuals will answer a clinical questionnaire and the International Physical Activity Questionnaire. The individual's clinical blood pressure will be checked (3 blood pressure checks on the arm with the highest value).

Anthropometry will be performed at the LIC and divided into assessment of total body mass, height and waist circumference.

The exercise test will be performed on a treadmill, with the Bruce Protocol, according to the Guidelines of the Brazilian Society of Cardiology. The test will be conducted in a specialized ICF/FUC room by a qualified professional in the presence of a cardiologist. Afterwards, the maximum oxygen consumption, respiratory equivalents and maximum heart rate will be lauded (prescription of aerobic exercises).

Step 2. The second visit will be held at the LIC, with the individual fasting for 12 hours for blood collection and biochemical analysis. After blood collection, a standardized snack will be offered and volunteers will be directed to a controlled room where they will lie for 10 minutes. The evaluation of arterial stiffness will be through the carotid-femoral pulse wave velocity (PWV), with Complior Analyze equipment®. The distance between the two points is measured by an infantometer and the data on blood pressure, height, total body mass and distance between the points of the carotid and femoral arteries are entered in the Complior Analyze software to calculate the PWV.

After analyzing the PWV, the volunteers will be tested for maximum strength of the lower limbs by testing a maximum repetition (1-RM). The test will be performed at the LIC in a specific environment for physical exercise (knee extension, knee flexion, leg pressure and plantar flexion exercises). A local warm-up will be performed with 10-12 repetitions and a load relative to 30% of the estimated weight for the 1-RM test and 2:2 cadence (concentric:eccentric), controlled by a metronome. After resting for 3-5 minutes, the 1-RM test will begin. The test will be interrupted to adjust the load when the individual performs more than 1-repetition or when he was unable to overcome the proposed load. When further attempts are required, a 5-minute rest period is allowed. The weight at which the individual performs only one repetition will be determined as 1-RM.

Step 3-4. To analyze the influence of the SNS on the FMD in response to physical exercise sessions, the α1-adrenergic blocking described in the literature will be used. Considering the interruption of the commercialization of the drug prazosin in Brazil, it will be replaced by its analogue doxazosin. Briefly, 90 minutes before starting the exercise protocol, individuals will be offered a capsule containing placebo (microcrystalline cellulose) or α1-adrenoreceptor blocker (Doxazosin 0.05 mg.kg-1 body weight) and will be instructed to lie down. A researcher collaborating in the group and blinded to the type of physical exercise, will be responsible for making the capsules available to the individual on the day of the session, according to previous randomization.

Evaluation of endothelial function: the evaluation of endothelial function will be performed by ultrasound using the FMD technique, as previously described. Initially, the speed of blood flow and the diameter of the brachial artery will be evaluated, simultaneously, in the volunteer's right arm, in a quiet, darkened room with controlled temperature (23-24°C) of the LIC, by a single qualified investigator and blinded to the condition. The initial blood pressure (left arm), resting heart rate, blood flow velocity and the diameter of the brachial artery will be evaluated after resting for 10-15 minutes in a supine position, with the subject's arm extended and positioned at an angle of ~40° of the trunk. The evaluation will take place 10 minutes before the exercise session, as well as 10-40-70 minutes after the exercise session.

To analyze the FMD of the brachial artery, individuals should be fasting for ≥6 hours, medicated for SAH. A rapid deflation cuff will be placed around the forearm 5 cm distal to the antecubital fossa and the image of the brachial artery will be obtained in the distal third of the arm in B-mode using a linear multi-frequency transducer (12MHz) connected to a high resolution Doppler Ultrasound system. The sample volume will be adjusted to cover the width of the vessel and an insonation angle of 60° will be used. Baseline diameters will be recorded for 1 minute, before the forearm cuff is inflated at 50 mmHg above the SBP, for 5 minutes. The recording of the images will be resumed 30 seconds before the deflation of the cuff and maintained for 3 minutes after deflation. The video signal of the Doppler Ultrasound will be recorded in real time by a USB video card and saved for offline analysis. The analysis of blood flow velocity and brachial artery diameter will be performed using edge detection and wall tracking software (CardiovasculareSuit™; Pisa, Italy). From the synchronized blood flow velocity data and the brachial artery diameter, the blood flow will be calculated at 30Hz. The FMD will be calculated as the percentage change in the peak diameter after deflating the cuff from the reference diameter (baseline).

Nervous system: the assessment of the ANS will be performed through the variability of heart rate and blood pressure, as already described in the literature. The data will be collected through the pressure wave acquisition system in a continuous and non-invasive way by the Finometer® system. For this, a cuffing will be installed on the middle finger (right hand) coupled to an analog-to-digital signal converter. The frequency of sampling the signals will be acquired continuously at 1000 Hz, after resting the individual (lying down for 10 minutes) and before the FMD analysis.

The collected data will be saved in the BeatsScope® and LabChart® software for analysis of blood pressure variability (BPV) histograms and pulse interval series (RR-interval) for spectral power analysis (heart rate variability, HRV). The pulse interval(PI) will be calculated as the difference between the start and end points of the cycle. The analysis of HRV and BPV in the time domain, such as the spectral composition (fast Fourier transform) will be performed using the CardioSeries® software (after removing transient and discrepant elements). The spectral bands for evaluation: very low frequency (VLF, 0.007-0.04Hz), low frequency (LF, 0.04-0.15Hz), high frequency (HF, 0.15-0.4Hz) and total power (TP, VLF+LF+HF). Spontaneous baroreflex sensitivity (SBE) will be inferred by the square root of (LF/HRV m2)/(LF/BPV m2).

The physical exercise sessions will be carried out in two visits, always in the afternoon (1:00 pm) and in random order for placebo or α1-adrenergic block. Moderate fasting (6 hours) will be required and sessions should have intervals of at least 5-7 days. The exercise sessions will be: aerobic, resistance and combined, previously published by our group.

The aerobic exercise session will be performed on a horizontal cycle ergometer. A warm-up will be performed (5 minutes), followed by 40 minutes with moderate intensity (60% HRreserve) and controlled by a heart rate monitor, as well as the subjective effort scale (Borg 6 to 20 points). Blood pressure, heart rate and the Borg scale will be assessed at the beginning of aerobic exercise and every 5 minutes until the end.

The resistance exercise session will be structured with knee extension, knee flexion, leg pressure and plantar flexion, in a station with guided weights, with 4x12 repetitions and 60% intensity of 1-RM; the cadence will be adjusted to 2:2 (concentric: eccentric) and controlled by a metronome. The rest between sets and exercises will be 90 seconds (total duration: 40 minutes). Blood pressure, heart rate and Borg scale will be recorded at the beginning and at the end of the 4th series of each exercise.

The combined exercise session will be structured with 20 minutes of resistance exercise + 20 minutes of aerobic exercise, as already described, except that the resistance exercises will have 2 sets of each exercise. As with other sessions, blood pressure, heart rate and the Borg scale will be assessed at the beginning and end of the second series of resistance exercise, as well as at the beginning and every 5 minutes of aerobic exercise up to 15 minutes after end of exercises.

Statistical analysis.

The normality of the data will be assessed by Shapiro-Wilk. Values will be presented as mean ± standard deviation or mediated and 95% CI, according to the distribution of variables. One-way ANOVA will be used for prior comparisons of baseline data between groups. The multivariate analysis of the data will be performed using the GEE for repeated measures with Bonferroni's post-hoc. The evaluation of possible correlations between variables will be performed using Pearson or Spearman tests. Statistical analysis: SPSS 24.0, p-value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of systemic arterial hypertension;
* Must be able to reality physical exercise.

Exclusion Criteria:

* Diabetes mellitus;
* Chronic renal failure;
* Body mass index ≥ 35kg/m2;
* Coronary artery disease;
* Heart failure;
* Use of beta-blocker;
* Uso of alpha-blocker;
* Smoker;
* Menopause (woman).

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-04-30 (Estimated); Primary Completion 2020-12-20 (Estimated); Study Completion 2021-12-23 (Estimated)

PRIMARY OUTCOMES:
Changes in the endothelial function of hypertensive individuals after a session of aerobic exercise, resistance exercise and combined exercise in α1-adrenoreceptor blocker and placebo condition. | Ten minutes before the exercise session and 10, 40 and 70 minutes after the exercise session.
  The method of assessing the flow-mediated dilation (FMD) of the brachial artery by ultrasonography is an indirect method to assess endothelial function. To analyze the FMD of the brachial artery a rapid deflation cuff will be placed around the forearm 5 cm distal to the antecubital fossa and the image of the brachial artery will be obtained in the distal third of the arm. Baseline diameters will be recorded for 1 minute, before the forearm cuff is inflated at 50 mmHg above the SBP, for 5 minutes. The recording of the images will be resumed 30 seconds before the deflation of the cuff and maintained for 3 minutes after deflation. The video signal of the Doppler Ultrasound will be recorded in real time by a USB video card and saved for offline analysis. The analysis of diameter will be performed using edge detection and wall tracking software. The FMD will be calculated as the percentage change in the peak diameter after deflating the cuff from the baseline diameter.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustavo Waclawovsky, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gimbrone MA Jr, Garcia-Cardena G. Endothelial Cell Dysfunction and the Pathobiology of Atherosclerosis. Circ Res. 2016 Feb 19;118(4):620-36. doi: 10.1161/CIRCRESAHA.115.306301. PMID 26892962
- [Background] Vanhoutte PM, Shimokawa H, Feletou M, Tang EH. Endothelial dysfunction and vascular disease - a 30th anniversary update. Acta Physiol (Oxf). 2017 Jan;219(1):22-96. doi: 10.1111/apha.12646. Epub 2016 Jan 25. PMID 26706498
- [Background] Iantorno M, Campia U, Di Daniele N, Nistico S, Forleo GB, Cardillo C, Tesauro M. Obesity, inflammation and endothelial dysfunction. J Biol Regul Homeost Agents. 2014 Apr-Jun;28(2):169-76. PMID 25001649
- [Background] Lind L. Lipids and endothelium-dependent vasodilation--a review. Lipids. 2002 Jan;37(1):1-15. doi: 10.1007/s11745-002-0858-6. PMID 11876256
- [Background] ESH/ESC Task Force for the Management of Arterial Hypertension. 2013 Practice guidelines for the management of arterial hypertension of the European Society of Hypertension (ESH) and the European Society of Cardiology (ESC): ESH/ESC Task Force for the Management of Arterial Hypertension. J Hypertens. 2013 Oct;31(10):1925-38. doi: 10.1097/HJH.0b013e328364ca4c. No abstract available. PMID 24107724
- [Background] Grassi G, Ram VS. Evidence for a critical role of the sympathetic nervous system in hypertension. J Am Soc Hypertens. 2016 May;10(5):457-66. doi: 10.1016/j.jash.2016.02.015. Epub 2016 Mar 4. PMID 27052349
- [Background] Ghorayeb N, Stein R, Daher DJ, Silveira ADD, Ritt LEF, Santos DFPD, Sierra APR, Herdy AH, Araujo CGS, Colombo CSSS, Kopiler DA, Lacerda FFR, Lazzoli JK, Matos LDNJ, Leitao MB, Francisco RC, Alo ROB, Timerman S, Carvalho T, Garcia TG. The Brazilian Society of Cardiology and Brazilian Society of Exercise and Sports Medicine Updated Guidelines for Sports and Exercise Cardiology - 2019. Arq Bras Cardiol. 2019 Mar;112(3):326-368. doi: 10.5935/abc.20190048. No abstract available. PMID 30916199
- [Background] Brandao AA, Amodeo C, Alcantara C, Barbosa E, Nobre F, Pinto F, Vilela-Martin JF, Bastos JM, Yugar-Toledo JC, Mota-Gomes MA, Neves MF, Malachias MV, Rodrigues MC, Passarelli O Junior, Jardim PC, Cunha PG, Povoa R, Fonseca T, Dias VP, Barroso WS, Oigman W. I Luso-Brazilian Positioning on Central Arterial Pressure. Arq Bras Cardiol. 2017 Feb;108(2):100-108. doi: 10.5935/abc.20170011. Epub 2017 Feb 13. No abstract available. PMID 28327876
- [Background] Thijssen DHJ, Bruno RM, van Mil ACCM, Holder SM, Faita F, Greyling A, Zock PL, Taddei S, Deanfield JE, Luscher T, Green DJ, Ghiadoni L. Expert consensus and evidence-based recommendations for the assessment of flow-mediated dilation in humans. Eur Heart J. 2019 Aug 7;40(30):2534-2547. doi: 10.1093/eurheartj/ehz350. PMID 31211361
- [Result] Soloviev MA, Kulakova NV, Semiglazova TA, Borodulina EV, Udut VV. Correction of endothelial dysfunction in patients with arterial hypertension. Bull Exp Biol Med. 2011 Jun;151(2):183-5. doi: 10.1007/s10517-011-1284-1. PMID 22238745
- [Result] Abebe W, Mozaffari M. Endothelial dysfunction in diabetes: potential application of circulating markers as advanced diagnostic and prognostic tools. EPMA J. 2010 Mar;1(1):32-45. doi: 10.1007/s13167-010-0012-7. Epub 2010 Mar 10. PMID 23199039
- [Result] Kublickiene K, Fu XD, Svedas E, Landgren BM, Genazzani AR, Simoncini T. Effects in postmenopausal women of estradiol and medroxyprogesterone alone and combined on resistance artery function and endothelial morphology and movement. J Clin Endocrinol Metab. 2008 May;93(5):1874-83. doi: 10.1210/jc.2007-2651. Epub 2008 Mar 4. PMID 18319309
- [Result] Pahkala K, Heinonen OJ, Simell O, Viikari JS, Ronnemaa T, Niinikoski H, Raitakari OT. Association of physical activity with vascular endothelial function and intima-media thickness. Circulation. 2011 Nov 1;124(18):1956-63. doi: 10.1161/CIRCULATIONAHA.111.043851. Epub 2011 Oct 3. PMID 21969011
- [Result] Green DJ, Dawson EA, Groenewoud HM, Jones H, Thijssen DH. Is flow-mediated dilation nitric oxide mediated?: A meta-analysis. Hypertension. 2014 Feb;63(2):376-82. doi: 10.1161/HYPERTENSIONAHA.113.02044. Epub 2013 Nov 25. PMID 24277765
- [Result] Dawson EA, Cable NT, Green DJ, Thijssen DHJ. Do acute effects of exercise on vascular function predict adaptation to training? Eur J Appl Physiol. 2018 Mar;118(3):523-530. doi: 10.1007/s00421-017-3724-8. Epub 2017 Dec 12. PMID 29234916
- [Result] Martinez DG, Nicolau JC, Lage RL, Toschi-Dias E, de Matos LD, Alves MJ, Trombetta IC, Dias da Silva VJ, Middlekauff HR, Negrao CE, Rondon MU. Effects of long-term exercise training on autonomic control in myocardial infarction patients. Hypertension. 2011 Dec;58(6):1049-56. doi: 10.1161/HYPERTENSIONAHA.111.176644. Epub 2011 Oct 24. PMID 22025377
- [Result] Hansen AH, Nyberg M, Bangsbo J, Saltin B, Hellsten Y. Exercise training alters the balance between vasoactive compounds in skeletal muscle of individuals with essential hypertension. Hypertension. 2011 Nov;58(5):943-9. doi: 10.1161/HYPERTENSIONAHA.111.176529. Epub 2011 Sep 6. PMID 21896936
- [Result] Nyberg M, Mortensen SP, Hellsten Y. Physical activity opposes the age-related increase in skeletal muscle and plasma endothelin-1 levels and normalizes plasma endothelin-1 levels in individuals with essential hypertension. Acta Physiol (Oxf). 2013 Mar;207(3):524-35. doi: 10.1111/apha.12048. Epub 2013 Jan 10. PMID 23227981
- [Result] Inaba Y, Chen JA, Bergmann SR. Prediction of future cardiovascular outcomes by flow-mediated vasodilatation of brachial artery: a meta-analysis. Int J Cardiovasc Imaging. 2010 Aug;26(6):631-40. doi: 10.1007/s10554-010-9616-1. Epub 2010 Mar 26. PMID 20339920
- [Result] Morishima T, Tsuchiya Y, Iemitsu M, Ochi E. High-intensity resistance exercise with low repetitions maintains endothelial function. Am J Physiol Heart Circ Physiol. 2018 Sep 1;315(3):H681-H686. doi: 10.1152/ajpheart.00281.2018. Epub 2018 Jun 1. PMID 29856651
- [Result] Atkinson CL, Lewis NC, Carter HH, Thijssen DH, Ainslie PN, Green DJ. Impact of sympathetic nervous system activity on post-exercise flow-mediated dilatation in humans. J Physiol. 2015 Dec 1;593(23):5145-56. doi: 10.1113/JP270946. Epub 2015 Nov 15. PMID 26437709
- [Result] Waclawovsky G, Umpierre D, Figueira FR, De Lima ES, Alegretti AP, Schneider L, Matte US, Rodrigues TC, Schaan BD. Exercise on Progenitor Cells in Healthy Subjects and Patients with Type 1 Diabetes. Med Sci Sports Exerc. 2016 Feb;48(2):190-9. doi: 10.1249/MSS.0000000000000764. PMID 26312614
- [Result] Torvik D, Madsbu HP. An open one-year comparison of doxazosin and prazosin for mild to moderate essential hypertension. Am J Cardiol. 1987 May 29;59(14):68G-72G. doi: 10.1016/0002-9149(87)90160-3. PMID 2884855
- [Result] Atala MM, Goulart A, Guerra GM, Mostarda C, Rodrigues B, Mello PR, Casarine DE, Irigoyen MC, Pereira AC, Consolim-Colombo FM. Arg16Gly and Gln27Glu beta2 adrenergic polymorphisms influence cardiac autonomic modulation and baroreflex sensitivity in healthy young Brazilians. Am J Transl Res. 2015 Jan 15;7(1):153-61. eCollection 2015. PMID 25755837
- [Derived] Waclawovsky G, Boll LFC, Neto SG, Irigoyen MCC, Lehnen AM. Effects of autonomic nervous system activation on endothelial function in response to acute exercise in hypertensive individuals: study protocol for a randomized double-blind study. Trials. 2021 Aug 19;22(1):548. doi: 10.1186/s13063-021-05516-x. PMID 34412668